CLINICAL TRIAL: NCT07325461
Title: Feasibility Study of Extended Wear Insulin Infusion Set Options During Home Use in People With Type 1 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-0023728
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; T1D; Tandem; t:slim X2; Tandem Mobi; automated insulin delivery; SteadiSet
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- t:slim X2 Users (Experimental): * t:slim X2 insulin pump with SteadiSet (43 inches) and an enhanced filling process (3 wear periods)
  * t:slim X2 with and SteadiSet (43 inches) with no side ports (3 wear periods)
  Interventions: Device: SteadiSet Infusion Set
- Mobi Users (Experimental): * Mobi Insulin Pump with SteadiSet (5 inches) and an enhanced filling process (3 wear periods)
  * Mobi Insulin Pump and SteadiSet (5 inches) (3 wear periods)
  Interventions: Device: SteadiSet Infusion Set

INTERVENTIONS:
Device: SteadiSet Infusion Set — Participants will use the SteadiSet Infusion set with an enhanced filling process for three wear periods and the Steadiset Infusion Set only for three wear periods.

SUMMARY:
This feasibility study is a prospective, single center, multi-arm study evaluating possible enhancements to the SteadiSet extended wear infusion set.

DETAILED DESCRIPTION:
All participants will use the SteadiSet insulin infusion set for 6 wear periods of up to 7 days each.

The 2 treatment arms are:

Existing t:slim X2 Users:

* t:slim X2 insulin pump with SteadiSet (43 inches) and an enhanced filling process (3 wear periods)
* t:slim X2 insulin pump with SteadiSet (43 inches) with no side ports (3 wear periods)

Existing Mobi Users:

* Mobi Insulin Pump with SteadiSet (5 inches) and an enhanced filling process (3 wear periods)
* Mobi Insulin Pump and SteadiSet (5 inches) (3 wear periods)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years old inclusive
* Generally in good health, as determined by the investigator
* Living in the United States with no plans to move outside the United States during the study
* Diagnosis of T1D for at least 12 months
* Currently using a Tandem pump
* Current Dexcom CGM user
* HbA1c <9.0% in the last 6 months.
* Willing to implement and adhere to pump alert/alarm settings on a study-provided pump as instructed during the study
* Willing to wear each investigational infusion set for up to 7 days during each of the wear periods in the study
* Willing to perform blood ketone and blood glucose (fingerstick) measurements as directed using provided ketone and blood glucose meters and strips
* If using Tandem Mobi, has a compatible cellular phone that can run the Tandem Mobi Mobile App
* BMI in the range 18-35 kg/m2, both inclusive
* Currently using one of the following insulins with no expectation of a need to change insulin type during the study:

  1. Humalog™ (or generic insulin lispro)
  2. NovoLog™ (or generic insulin aspart)
* Willing to change insulin cartridge every 48-72 hours, as recommended by patient's healthcare provider during the study
* Has the ability to understand and comply with protocol procedures and to provide informed consent

Exclusion Criteria:

* Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
* Female subject is pregnant, planning to become pregnant, or not using adequate method of contraception
* Episodes of severe hypoglycemia in the last 6 months resulting in:

  1. Medical Assistance (i.e., paramedics, hospital evaluation or hospitalization)
  2. Loss of consciousness
  3. Seizures
* One or more episodes of diabetic ketoacidosis (DKA) in the last 6 months requiring hospitalization
* Currently on a ketogenic or low-carbohydrate diet of less than 60 grams of carbohydrates per day, or intending to begin one during the study period
* Known history of any of the following conditions:

  1. Cushing's Disease
  2. Adrenal insufficiency
  3. Pancreatic islet cell tumor
  4. Insulinoma
  5. Lipodystrophy
  6. Extensive lipohypertrophy, as assessed by the investigator
* Undergoing treatment with systemic oral or intravenous corticosteroids, at or within the last 8 weeks from screening. Inhaled glucocorticoids are allowed.
* Significant history of any of the following, that in the opinion of the investigator would compromise safety or successful study participation:

  1. Alcoholism
  2. Drug abuse
* Significant acute or chronic illness, that in the opinion of the investigator might interfere with safety or integrity of study results
* Current participation in another clinical drug or device study
* Immediate family member (spouse, biological or legal guardian, child, sibling, parent) who is a study site personnel directly affiliated with this study or who is an employee of Tandem Diabetes Care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
7 Day Survival of Infusion Set for Primary Outcome Measure | 6 weeks
  7-day infusion set survival for primary outcome reasons as defined in the protocol (Hyperglycemia and failure to respond to boluses, Hyperglycemia with ketones >1.0 mmol/L, or Investigator advised)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No